CLINICAL TRIAL: NCT06688279
Title: Effects of Plyometric Exercises on Strength, Power and Dynamic Balance in Female Fast Bowlers
Brief Title: Effects of Plyometric Exercises in Female Fast Bowlers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0423
Record Dates: First submitted 2024-10-15; First posted 2024-11-14 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Plyometric Exercises; Strength; Dynamic Balance; Power
Keywords: Plyometric Exercises; Strength; dynamic balance; power
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: There will be two groups included in this study. Group A: It will receive 8 weeks of upper and lower body plyometric exercises protocol.
  Group B: It will receive 8 weeks of standard exercises protocol.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plyometric exercises protocol (Experimental): 14 female fast bowlers will receive 8 weeks of upper and lower body plyometric exercises protocol. The session will last for 60 minutes and 3 times per week. 5 minutes warm up with dynamic stretching and 5 minutes cool down period with static stretching and 1-minute rest period is there between each exercise and each repetition and 3-5 minute for each set (total 3 sets).
  Following Plyometrics would be performed.
  1. Plyo Pushup.
  2. Chest Pass.
  3. Overhead Throw.
  4. Squat jump.
  5. Plyo Step-up.
  6. Cone jumps.
  7. Med Ball drop.
  8. Kneeling Squat jump.
  9. Lateral jump over hurdle.
  10. Overhead throw.
  11. Under hand throws.
  12. Dynamic Rotational Chest pass.
  13. Overhead throw with step. Vertical jump test for lower extremity strength, 3-Hop test for lower extremity power and Star excursion balance test for dynamic balanceis performed at the start of exercise protocol and in the end i.e. Pre and post test.
  Interventions: Other: Plyometric Exercise
- Standard exercises protocol (Experimental): 14 female fast bowlers will receive their standard exercise protocol. The session will last for 60 minutes and 3 times per week.
  Following exercises would be performed.
  * Push ups.
  * Sit ups.
  * Lunges
  * 500 m running.
  * Squats Vertical jump test for lower extremity strength, 3-Hop test for lower extremity power and Star excursion balance test for dynamic balanceis performed at the start of exercise protocol and in the end i.e. Pre and post test.
  Interventions: Other: Standard exercises protocol

INTERVENTIONS:
Other: Plyometric Exercise — . The session will last for 60 minutes and 3 times per week. 5 minutes warm up with dynamic stretching and 5 minutes cool down period with static stretching and 1-minute rest period is there between each exercise and each repetition and 3-5 minute for each set (total 3 sets).
  Following Plyometrics would be performed.
  1. Plyo Pushup.
  2. Chest Pass.
  3. Overhead Throw.
  4. Squat jump.
  5. Plyo Step-up.
  6. Cone jumps.
  7. Med Ball drop.
  8. Kneeling Squat jump.
  9. Lateral jump over hurdle.
  10. Overhead throw.
  11. Under hand throws.
  12. Dynamic Rotational Chest pass.
  13. Overhead throw with step. Vertical jump test for lower extremity strength, 3-Hop test for lower extremity power and Star excursion balance test for dynamic balanceis performed at the start of exercise protocol and in the end i.e. Pre and post test.
  Arms: Plyometric exercises protocol
Other: Standard exercises protocol — The session will last for 60 minutes and 3 times per week. Following exercises would be performed.
  * Push ups.
  * Sit ups.
  * Lunges
  * 500 m running.
  * Squats Vertical jump test for lower extremity strength, 3-Hop test for lower extremity power and Star excursion balance test for dynamic balanceis performed at the start of exercise protocol and in the end i.e. Pre and post test.
  Arms: Standard exercises protocol

SUMMARY:
Cricket is one of the most popular team sports in the world. Bowling action is an extremely skilled activity that has been developed over many years of practice. Physiological variables and an imbalance between the agonist and antagonist muscle groups are important risk factors for development in high skill bowlers.

Exercises known as plyometric training use explosive motions to build muscle mass and improve aspects of physical fitness. Ballistic six plyometric exercises have been shown to improve performance in medium-paced cricket bowlers by increasing bowling velocity.This randomized controlled trial will be conducted in Pakistan Sports Board Lahore. This study will be completed in 10 months after the approval of synopsis. Non-probability convenient sampling technique will be used. Inclusion criteria will include female fast bowlers with age group between19 to 27years who are active team members of their respective leagues without the presence of injuries and whose composite score will be greater than 75 on star excursion balance scale will be included. Any participant post-elbow or shoulder surgery within one year of the study's pre-test or presenting with a history of elbow or shoulder injury or pain within one year of the study's pre-test will be excluded. The study will be conducted in two groups. Group A (14 players) will receive 8 weeks of upper and lower body plyometric exercises protocol. The session will last for 60 minutes and 3 times per week.10-15 mints warm up before plyometric exercises and 1-minute rest period is there between each exercise and each repetition and 3-5 minute for each set. Group B (14 players) will receive their standard exercise protocol. The session will last for 60 minutes and 3 times per week. Vertical jump test for lower extremity strength, 3-Hop test for lower extremity power and Star excursion balance test for dynamic balance is performed at the start of exercise protocol and in the end. After data collection data will be analyzed using statistical package for social sciences SPSS version 21.

DETAILED DESCRIPTION:
Cricket is one of the most popular team sports in the world. Bowling action is an extremely skilled activity that has been developed over many years of practice. Physiological variables and an imbalance between the agonist and antagonist muscle groups are important risk factors for development in high skill bowlers. Physical improvements have a significant impact on team sports since players undertake several explosive movements during the game such as hitting, jumping, turning, sprinting, and altering speed and direction.Exercises known as plyometric training use explosive motions to build muscle mass and improve aspects of physical fitness. Ballistic six plyometric exercises have been shown to improve performance in medium-paced cricket bowlers by increasing bowling velocity. Plyometric exercises have emerged as a catalyst for transformative improvements in athletic performance.Our exploration goes beyond the realms of traditional training, aiming to unravel the intricacies of how plyometrics can be harnessed to sculpt not only strength and power but also dynamic balance in these athletes.

This randomized controlled trial will be conducted in Pakistan Sports Board Lahore. This study will be completed in 10 months after the approval of synopsis. Non-probability convenient sampling technique will be used. Sample size with 20% attrition rate is 28 which is calculated using G-Power. Inclusion criteria will include female fast bowlers with age group between19 to 27years who are active team members of their respective leagues without the presence of injuries and whose composite score will be greater than 75 on star excursion balance scale will be included. Any participant post-elbow or shoulder surgery within one year of the study's pre-test or presenting with a history of elbow or shoulder injury or pain within one year of the study's pre-test will be excluded.The study will be conducted in two groups. Group A (14 players) will receive 8 weeks of upper and lower body plyometric exercises protocol. The session will last for 60 minutes and 3 times per week.10-15 mints warm up before plyometric exercises and 1-minute rest period is there between each exercise and each repetition and 3-5 minute for each set. Group B (14 players) will receive their standard exercise protocol. The session will last for 60 minutes and 3 times per week. Vertical jump test for lower extremity strength, 3-Hop test for lower extremity power and Star excursion balance test for dynamic balance is performed at the start of exercise protocol and in the end. After data collection data will be analyzed using statistical package for social sciences SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Patient between age of 19 to 28 years
* Female fast bowlers.
* Active team members of their respective leagues.
* Healthy, without the presence of injuries.
* Whose composite score will be greater than 75 on star excursion balance scale.

Exclusion Criteria:

* Femles with Injury.
* History of elbow or shoulder injury or pain within one year of the study's pre-test will be excluded.

Ages: 19 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Vertical jump test for lower extremity strength | 8 weeks
  The knee angle was 90 degrees at the start of the vertical jump. In order to do a vertical leap, subjects had to push upward while maintaining a straight leg throughout to avoid falling. The patients were standing when the countermovement leap started, standing erect and rapidly descending to a 90-degree angle at the knees before launching off. The participants may do as they pleased. In the third test, they will use their hands to jump. One minute of break was allowed in between each of the three trials, with the top values for every leap that will be applied in later examinations. It is the most valid and reliable test for lower extremity strength
3-Hop test for lower extremity power | 8 week
  The triple hop test is frequently used to evaluate a lower limb's functional strength, power, or neuromuscular control the evaluation of a person's capacity to minimize movement by jumping and landing on one foot without taking a step.
  Starting with their toe on the starting line, the athlete should stand on the assigned test leg. When the competitor is prepared, they will utilize the assigned leg; make three consecutive, maximum jumps forward. The tester will calculate the distance jumped from the starting line until the subject's heel touches down after making their third leap. When doing a single-leg horizontal hop, the upper limbs move. Testing is not restricted, although participants are told to adhere to the landing on the last hop. The athlete will not change after landing the landing foot or to let the supporting foot of the opposing foot touch the ground. One step must be finished in a single second. Athletes were limited to three repetitions. There should be a 30-second bre
Star excursion balance test for dynamic balance | 8 weeks
  The player remained on 1 leg in the focal point of a matrix, with the most distal part of the extraordinary toe at the beginning line. While keeping up with single-leg position, the player was approached to reach with the free limb in the anterior, postero-medial, and postero-lateral headings in relation to the position foot. The maximal reach distance was estimated by denoting the measuring tape with erasable ink where the most distal some portion of the foot came to. The preliminary was disposed of and rehashed if the player neglected to keep up with unilateral position, lifted or moved the position foot from the network, landed with the reach foot or neglected to return the reach foot to the beginning position. Standing on the opposite leg, the procedure was carried out once more. For the purpose of analyzing the reach distance in each direction, the three highest trials for each reach direction were used. Likewise, the best reach at distance from every heading was added to yield

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pardos-Mainer E, Lozano D, Torrontegui-Duarte M, Carton-Llorente A, Roso-Moliner A. Effects of Strength vs. Plyometric Training Programs on Vertical Jumping, Linear Sprint and Change of Direction Speed Performance in Female Soccer Players: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jan 6;18(2):401. doi: 10.3390/ijerph18020401. PMID 33419178
- [Background] Makhlouf I, Chaouachi A, Chaouachi M, Ben Othman A, Granacher U, Behm DG. Combination of Agility and Plyometric Training Provides Similar Training Benefits as Combined Balance and Plyometric Training in Young Soccer Players. Front Physiol. 2018 Nov 13;9:1611. doi: 10.3389/fphys.2018.01611. eCollection 2018. PMID 30483158
- [Background] Werfelli H, Hammami R, Selmi MA, Selmi W, Gabrilo G, Clark CCT, Duncan M, Sekulic D, Granacher U, Rebai H. Acute Effects of Different Plyometric and Strength Exercises on Balance Performance in Youth Weightlifters. Front Physiol. 2021 Sep 14;12:716981. doi: 10.3389/fphys.2021.716981. eCollection 2021. PMID 34594236
- [Background] Lu Z, Zhou L, Gong W, Chuang S, Wang S, Guo Z, Bao D, Zhang L, Zhou J. The Effect of 6-Week Combined Balance and Plyometric Training on Dynamic Balance and Quickness Performance of Elite Badminton Players. Int J Environ Res Public Health. 2022 Jan 30;19(3):1605. doi: 10.3390/ijerph19031605. PMID 35162627
- [Background] Caron KE, Burr JF, Power GA. The Effect of a Stretch-Shortening Cycle on Muscle Activation and Muscle Oxygen Consumption: A Study of History-Dependence. J Strength Cond Res. 2020 Nov;34(11):3139-3148. doi: 10.1519/JSC.0000000000003815. PMID 33105364
- See also: The Effect of a Stretch-Shortening Cycle on Muscle Activation and Muscle Oxygen Consumption: A Study of History-Dependence — https://pubmed.ncbi.nlm.nih.gov/33105364
- See also: The Effect of 6-Week Combined Balance and Plyometric Training on Dynamic Balance and Quickness Performance of Elite Badminton Players — https://pubmed.ncbi.nlm.nih.gov/35162627
- See also: Acute Effects of Different Plyometric and Strength Exercises on Balance Performance in Youth Weightlifters — https://pubmed.ncbi.nlm.nih.gov/34594236
- See also: Effects of Strength vs. Plyometric Training Programs on Vertical Jumping, Linear Sprint and Change of Direction Speed Performance in Female Soccer Players: A Systematic Review and Meta-Analysis — https://pubmed.ncbi.nlm.nih.gov/33419178